CLINICAL TRIAL: NCT03966898
Title: A Phase III Study to Evaluate Efficacy and Safety of SHR6390 in Combination With Letrozole or Anastrozole Versus Placebo in Combination With Letrozole or Anastrozole in Patients With HR Positive and HER2 Negative Recurrent/Metastatic Breast Cancer
Brief Title: A Study of SHR6390 in Combination With Letrozole or Anastrozole in Patients With HR Positive and HER2 Negative Advanced Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR6390-III-302
Record Dates: First submitted 2019-05-21; First posted 2019-05-29 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2020-06

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Letrozole; Anastrozole

STUDY DESIGN:
Intervention Model Description: SHR6390 in combination with Letrozole or Anastrozole versus placebo in combination with Letrozole or Anastrozole
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR6390, Letrozole or Anastrozole (Experimental): SHR6390, Letrozole or Anastrozole
  Interventions: Drug: SHR6390 Tablets; Drug: Letrozole or Anastrozole Tablets
- Placebo, Letrozole or Anastrozole (Placebo Comparator): Placebo, Letrozole or Anastrozole
  Interventions: Drug: Placebo Tablets; Drug: Letrozole or Anastrozole Tablets

INTERVENTIONS:
Drug: SHR6390 Tablets — SHR6390 Tablets
  Arms: SHR6390, Letrozole or Anastrozole
Drug: Placebo Tablets — Placebo Tablets
  Arms: Placebo, Letrozole or Anastrozole
Drug: Letrozole or Anastrozole Tablets — Letrozole or Anastrozole Tablets

SUMMARY:
This is a phase III clinical trial to evaluate the efficacy and safety of SHR6390 in combination with Letrozole or Anastrozole versus placebo in combination with Letrozole or Anastrozole in Patients who have HR positive and HER2 negative recurrent/metastatic breast cancer and have not received systemic anticancer therapy are eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Has the pathologically-confirmed diagnosis of locally recurrent or metastatic, hormone-receptor positive, HER2 negative Breast Cancer.
2. Age: 18 - 75 years old
3. No prior systemic anti-cancer therapy for advanced HR+ disease.
4. Eastern Cooperative Oncology Group [ECOG] 0-1

Exclusion Criteria:

1. Patients who received prior treatment with any CDK4/6 inhibitor.
2. Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), or ventricular arrhythmia which need medical intervention.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed PFS | Every 8 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, Up to approximately 24 months.
  Investigator-assessed Progression Free Survival

SECONDARY OUTCOMES:
Progression-free Survival (PFS) per RECIST 1.1 | Up to approximately 24 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first.
OS | up to 2 years
  Overall Survival
ORR | Up to approximately 24 months
  Objective Response Rate
DoR | Up to approximately 24 months
  Duration of Objective Response
CBR | Up to approximately 24 months
  Clinical Benefit rate
Number of Participants With adverse events (AEs) and serious adverse events (SAEs) Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0 | Up to approximately 24 months
  Number of Participants With adverse events and serious adverse events Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0

OTHER OUTCOMES:
Ctrough | Up to 4 weeks
  To explore the pharmacokinetic characteristics of SHR6390 population and the influencing factors

CONTACTS AND LOCATIONS:
Locations (1):
- Nayima Bayaxi, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong J, Chen T, Ouyang L, Du N, Li A, Zhou Z, Zhang H, Xia Z, Meng J. Cost-effectiveness comparison of dalpiciclib and abemaciclib combined with an aromatase inhibitor as first-line treatment for HR+/HER2- advanced breast cancer. Expert Rev Pharmacoecon Outcomes Res. 2024 Apr;24(4):559-566. doi: 10.1080/14737167.2024.2330542. Epub 2024 Mar 20. PMID 38470447
- [Derived] Zhang P, Zhang Q, Tong Z, Sun T, Li W, Ouyang Q, Hu X, Cheng Y, Yan M, Pan Y, Teng Y, Yan X, Wang Y, Xie W, Zeng X, Wang X, Hu C, Geng C, Zhang H, Li W, Wu X, Zhong J, Xu J, Shi Y, Wei W, Bayaxi N, Zhu X, Xu B. Dalpiciclib plus letrozole or anastrozole versus placebo plus letrozole or anastrozole as first-line treatment in patients with hormone receptor-positive, HER2-negative advanced breast cancer (DAWNA-2): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2023 Jun;24(6):646-657. doi: 10.1016/S1470-2045(23)00172-9. Epub 2023 May 11. PMID 37182538